CLINICAL TRIAL: NCT00793884
Title: Emory Latino Diabetes Education Program
Acronym: ELDEP
Status: Suspended | Type: Observational
Why Stopped: Enrollment and study activities are temporarily suspended pending additional funding.
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry); Eli Lilly and Company (Industry); Takeda (Industry); Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Other Study IDs: IRB00013340
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Diabetes
Keywords: Diabetes; Latino population
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Diabetes Education: Latino individuals with diabetes who are attending the Emory Latino Diabetes Education Program (ELDEP) will be followed in order to collect outcomes on clinical measurements. The class curriculum follows the American Association of Diabetes Educators (AADE) seven self-care behaviors: healthy eating, being active, monitoring, medication use, problem-solving and healthy coping. Program participants attend an initial 3 hour diabetes education class conducted in Spanish and then are invited to return to monthly follow-up sessions covering topics of meal planning, exercise, medications and complications. The follow-up sessions include activities such as dance lessons, cooking demonstrations, and sharing.

SUMMARY:
Latinos with diabetes who are attending the Emory Latino Diabetes education program will be approached about consenting to have clinical measurements collected to assess changes between baseline and monthly follow up sessions. The no-cost educational sessions follow the self-care behavior curriculum of the American Association of Diabetes Educators (AADE).

DETAILED DESCRIPTION:
Latinos represent the largest minority group in the United States with a population of 35 million or 12.5%. National surveys indicate that the prevalence of type 2 diabetes is 1.9 times higher in Latinos than non-whites, and that approximately 24% percent of Latinos over the age of 45 years have diabetes. In Georgia, Latinos make up approximately 6.5% of the population. During 1990 and 2000, the prevalence of diabetes in Fulton and Dekalb counties, two of the most populated areas in Georgia and the Atlanta metropolitan area increased by 30%. Language and cultural barriers represent the two most important obstacles in educating and improving the care of Latino patients with diabetes. Less than 5% of physicians, 2% of nurses, and 2.5% of dentists in the US speak Spanish.

The Emory Latino Diabetes education program has been in existence since December 2005. This program aims to deliver diabetes education in Spanish to the underserved Latino community in Metro Atlanta. Program participants attend an initial 3 hour diabetes education class in Spanish. The class curriculum follows the American Association of Diabetes Educators (AADE) seven self-care behaviors: healthy eating, being active, monitoring, medication use, problem-solving and healthy coping. Participants are invited to return to a follow-up session within 6 months. Follow-up sessions are held in the late afternoon. These sessions are discussion-based and include an activity such as salsa lessons and cooking demonstrations. Diabetes education classes and follow-up sessions are offered at Grady Memorial Hospital (Diabetes Clinic, International Medical Center), Grady North Dekalb Clinic (Chamblee), and North Fulton Regional Hospital.

Participants complete a questionnaire assessing behaviors and social and demographic characteristics of the Latino community being served. Hemoglobin A1C, blood pressure, weight, body mass index (BMI) and waist circumference will be measured at the beginning of each class. This study will analyze and publish data collected from individuals who are attending the educational sessions. Additionally, the researchers will collect retrospective data from past participants in the program.

ELIGIBILITY:
Inclusion Criteria:

* spanish speaking patients with diabetes

Exclusion Criteria:

* under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spanish speaking patients with Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2008-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Social and Demographic Characteristics | 5 years
  One aim of this study is to describe the social and demographic characteristics of the Latino population with diabetes mellitus in Georgia. Participants will complete a qualitative demographic survey including questions regarding medical care received, physical activity, medications taken and blood sugar monitoring habits.

SECONDARY OUTCOMES:
Barriers to Health Care | 5 years
  To examine barriers to health care among Latinos with Diabetes in the population served participants will be asked qualitative questions about what type of health insurance they have and if they have a physician that they see.
Change in Blood Glucose Level | Baseline, Montly Follow-up Visits (up to 5 years)
  Blood glucose levels are measured in milligrams of glucose per deciliter of blood (mg/dL). Normal fasting levels are between 70 and 99 mg/dL and diabetes is indicated when fasting glucose levels are greater than 125 mg/dL.
Change in Hemoglobin A1C | Baseline, Montly Follow-up Visits (up to 5 years)
  The hemoglobin A1c test result is reported as a percentage. Higher percentages indicate higher blood glucose levels in the previous three months. A normal HbA1c level is below 5.7 percent.
Change in Waist Circumference | Baseline, Montly Follow-up Visits (up to 5 years)
  Waist circumference is measured in centimeters (cm).
Change in Body Mass Index (BMI) | Baseline, Montly Follow-up Visits (up to 5 years)
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters.
Change in Systolic Blood Pressure | Baseline, Montly Follow-up Visits (up to 5 years)
  Blood pressure will be measured using blood pressure monitor. Normal systolic blood pressure is less than 120 millimeter of mercury (mm/Hg) and high blood pressure is typically diagnosed at measurements of 130 mm/Hg and higher.
Change in Diastolic Blood Pressure | Baseline, Montly Follow-up Visits (up to 5 years)
  Blood pressure will be measured using blood pressure monitor. Normal diastolic blood pressure is less than 80 mm/Hg and high blood pressure is typically diagnosed at measurements of 80 mm/Hg and higher.

CONTACTS AND LOCATIONS:
Overall Officials: Ina Flores, MS, RN, CDE, LD, Study Director — Emory University; Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Emory University School of Medicine, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No